CLINICAL TRIAL: NCT00426127
Title: Phase II Trial of Docetaxel and Liposomal Doxorubicin (Doxil) Chemotherapy Combined With Enoxaparin in Patients With Advanced Pancreatic Cancer
Brief Title: Docetaxel and Liposomal Doxorubicin Chemotherapy With Enoxaparin in Patients With Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate number of eligible patients
Sponsor: University of Iowa (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Daniel Berg, Principal Investigator, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200511721
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic; Docetaxel; Doxorubicin; Enoxaparin
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Docetaxel; liposomal doxorubicin; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel and Liposomal Doxorubicin Combined with Enoxaparin (Experimental): Docetaxel 75 mg/m^2 + Doxil 30 mg/m^2 + Enoxaparin 1.5 mg/kg
  Interventions: Drug: Docetaxel; Drug: Liposomal Doxorubicin; Drug: Enoxaparin

INTERVENTIONS:
Drug: Docetaxel
  Other Names: Taxotere
Drug: Liposomal Doxorubicin
  Other Names: caelyx
Drug: Enoxaparin
  Other Names: Lovenox

SUMMARY:
The purpose of this study is to assess the effects of the treatment combination of the commercially available chemotherapy drugs, docetaxel and liposomal doxorubicin, and a blood thinner Enoxaparin on pancreatic cancer. The main goal of the study is to find out if this combination chemotherapy and enoxaparin increases the number of individuals whose tumors shrink.

DETAILED DESCRIPTION:
The objective of the study is to determine the safety and efficacy of the combination of docetaxel and liposomal doxorubicin chemotherapy combined with enoxaparin in patients with advanced pancreatic cancer.

Docetaxel (TAXOTERE) belongs to the group of anticancer drugs called mitotic inhibitors. Liposomal doxorubicin (Doxil) is an anthracycline, and is thought to prevent nucleic acid synthesis that is needed to make DNA. Enoxaparin (Lovenox) is an anticoagulant. We are interested in combining chemotherapy with the blood thinner enoxaparin because there is a scientific link between blood clotting and malignancy.

This research is being done to improve on currently available chemotherapy treatments for advanced pancreatic cancer. The main goal of the study is to find out if this combination chemotherapy and enoxaparin increases the number of individuals whose tumors shrink. Another purpose of this study is to find out how this study treatment effects blood clotting levels in individuals. We will also determine the incidence of elevated D-dimer and the effect of this regimen on the level of D-dimer, and collect safety data on this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed pancreatic carcinoma, with at least one lesion measurable by CT scan with a longest diameter of > 10mm, (other than bone) that has either not been previously irradiated, or if previously irradiated, has demonstrated progression since the radiation therapy based on RECIST criteria.
* Locally-advanced unresectable disease or be ineligible for neo-adjuvant therapy (Stage III disease, unresectable and medically unfit for neo-adjuvant treatment or decline chemo radiation treatment) or have metastatic disease.
* 18 years of age or greater. Female patients with child-bearing potential must have a negative pregnancy test at screening. All patients of reproductive potential must agree to practice effective contraception in order to participate in this study for duration of treatment and for 3 months post.
* WBC >3000 cells/mm3 with segments over 1800, hemoglobin >10 g/dl, platelets >150,000 cells/mm3, creatinine <1.5 mg/dl.
* Hepatic function: Total Bilirubin </= ULN. AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values (AST or ALT) should be used.
* ECOG performance status of </= 2 and an expected survival of at least 3 months.
* Stable neurological status without clinical evidence of CNS metastases and/or stroke. Peripheral neuropathy must be </= Grade 1.

Exclusion Criteria:

* Chemotherapy or radiation therapy within the preceding 4 weeks. Patients must never have had docetaxel or liposomal or regular doxorubicin.
* Spinal/epidural anesthesia and/or catheters for pain management
* New York Heart Association (NYHA) class III or IV congestive heart failure
* Evidence of duodenal erosion from the cancer.
* Heparin or coumadin at the time of enrollment, with the exception of low dose coumadin (1 mg/day or less) administered prophylactically and/or heparin for maintenance of in-dwelling lines or ports.
* Acute DVT or PE on initial evaluation
* History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* Pregnant or breast feeding
* Undergone a major surgical procedure, open biopsy, or major traumatic injury less than 4 weeks prior to study entry. Fine needle aspirations or venous access devices are allowed if placed > 7 days before study treatment begins.
* Presence of active or suspected acute or chronic uncontrolled infection, including abscess or fistula
* HIV positive
* History of another malignancy within 5 years prior to study entry, except curatively treated basal cell skin cancer or cervical cancer in situ
* Medical or psychiatric illness that would preclude study or informed consent and/or history of noncompliance to medical regimens or inability or unwillingness to return for all scheduled visits
* Enoxaparin is contraindicated in patients with active major bleeding or who are at high risk for bleeding, in patients with thrombocytopenia associated with a positive in vitro test for anti-platelet antibody in the presence of enoxaparin sodium, or in patients with hypersensitivity to enoxaparin sodium. Patients with known hypersensitivity to heparin or pork products should not be treated with enoxaparin injection or any of its constituents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Berg, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for Holden Comprehensive Cancer Center at University of Iowa — http://www.uihealthcare.com/depts/cancercenter/index.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel and Liposomal Doxorubicin Combined With Enoxaparin: Docetaxel 75 mg/m^2 + Doxil 30 mg/m^2 + Enoxaparin 1.5 mg/kg
  Docetaxel
  Liposomal Doxorubicin
  Enoxaparin
Period: Overall Study
Arm/Group | Docetaxel and Liposomal Doxorubicin Combined With Enoxaparin
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Removed due to disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel and Liposomal Doxorubicin Combined With Enoxaparin
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants] — Population: Participants who received study treatment
  Participants
    <=18 years | 0
    Between 18 and 65 years | 1
    >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] — Population: Participants who received study treatment
  Years | 61.8 [58.2 to 65.5]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants who received study treatment
  Participants
    Female | 2
    Male | 0
Region of Enrollment [Number; unit: participants] — Population: Participants who received study treatment
  participants
    United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Measured by CT Scans After Each Set of 3 Cycles of Chemotherapy
Time Frame: 9 weeks
Population: One participant underwent 3 cycles of therapy and progressed as assessed by CT.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel and Liposomal Doxorubicin Combined With Enoxaparin
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Number of Blood Draws With Incidence of Elevated D-Dimer Measured by Drawing D-Dimer Levels Every Cycle
Description: Incidence of elevated D-Dimer was defined as >.50 as drawn every cycle. Incidence of elevated D-Dimer was tested to determine safety and efficacy of the treatment regimen on patients with advanced pancreatic cancer.
Time Frame: 3 weeks
Population: 2 patients received at least one cycle of treatment and underwent blood draws testing D-Dimer levels
Measure: Number; unit: Blood draw
Arm/Group | Docetaxel and Liposomal Doxorubicin Combined With Enoxaparin
Number analyzed (Participants) | 2
Blood draw
  Incidences within normal range D-Dimer <.50 | 3
  Incidence with elevated D-Dimer >.50 | 1

3. Secondary Outcome: Safety and Effect of Chemo Regimen on D-Dimer Measured by Drawing D-Dimer Levels Every Cycle
Time Frame: 3 weeks
Population: There was no analysis done
Arm/Group | Docetaxel and Liposomal Doxorubicin Combined With Enoxaparin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All patients underwent a history and physical examination every 3 weeks during the therapy.
Arm/Group | Docetaxel and Liposomal Doxorubicin Combined With Enoxaparin
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Liposomal Doxorubicin Combined With Enoxaparin (N=2)
Disease progression (General disorders) | 1 (1) — Patient had expired due to rapidly progressive disease within 30 days of last dose of study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Liposomal Doxorubicin Combined With Enoxaparin (N=2)
Weight loss (Investigations) | 1 (1)
Neutropenia (Immune system disorders) | 1 (1)
Decreased white blood cell count (Investigations) | 1 (1)
Decreased hemoglobin (Investigations) | 1 (1)
Decreased calcium (Investigations) | 1 (1)
Decreased albumin (Investigations) | 1 (1)
Increased alk phosphatase (Investigations) | 1 (1)
Decreased sodium, intermittent (Investigations) | 1 (1)
Decreased phosphate (Investigations) | 1 (1)
Ascites, worsening recurrent (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pedal edema (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Oral thrush (Infections and infestations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Difficulty sleeping (Psychiatric disorders) | 1 (2)
Injection site pain (General disorders) | 1 (1)
Hand foot syndrome (red feet) (General disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 2 (2)
Oral mucositis (Gastrointestinal disorders) | 2 (3)
Itching (General disorders) | 1 (1)
Sensory neuropathy (General disorders) | 1 (1) — "Hot tongue"
Nasal sores (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Taste disturbance (Nervous system disorders) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Ecchymosis, injection site (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Rash of underarm
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Chills (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study closed early due to slow accrual. No analysis done, 2 subjects received study treatment. Both subjects went off study due to progression and complications from cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes